CLINICAL TRIAL: NCT07344090
Title: PREMARKET INVESTIGATION ON THE USE OF A DIGITAL DECISION-MAKING AID AIMED AT IMPROVING THE APPROPRIATENESS AND ADHERENCE TO THERAPY FOR THE MANAGEMENT OF FEVER AND ACUTE PAIN IN PATIENTS BETWEEN 3 MONTHS AND 1 DAY AND 5 YEARS OF AGE
Brief Title: USING A DECISION-MAKING SYSTEM TO SUPPORT THE MANAGEMENT OF FEVER AND ACUTE PAIN IN CHILDREN
Acronym: FEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qwince Innovation S.r.l. (Industry)
Collaborators: Consorzio per Valutazioni Biologiche e Farmacologiche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-CE-29153; EUDAMED Number 25-10-054835 (Other: European Commission)
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fever, Acute Pain
Keywords: fever, acute pain, pediatrics
MeSH Terms: conditions — Fever; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): After signing the informed consent, the patient and caregiver will be enrolled in the study and registered in the Puntofarma® system, resulting in the issuance of a unique code. No personal data of the patient and/or caregiver will be recorded on the device.
  At the same time, a PIN code will be issued for each enrolled patient, allowing the caregiver to register in the digital application and begin using the algorithm from their mobile/digital device.
  Caregivers will be required to enter the necessary information into the application so that the algorithm can calculate the recommended dose of paracetamol. The application, which can be downloaded to a mobile phone, is used to verify adherence to the antipyretic therapy suggested by the algorithm and based on the guidelines for the management of fever and acute pain in children.
  Interventions: Device: Puntofarma® FEVER

INTERVENTIONS:
Device: Puntofarma® FEVER — Puntofarma® is a software-based medical device, which the manufacturer intends to use in standalone mode, with the aim of improving prevention, monitoring, and patient care processes.
  In the context of the FEVER clinical trial, it is designed to:
  * acquire and organize pediatric patient health information (measurements, parameters);
  * assist caregivers/parents in managing fever/acute pain, including through alarms and reminders;
  * create a communication channel between caregivers/parents and healthcare professionals.
  The clinically relevant features of Puntofarma® for the FEVER study are as follows:
  * collect data regarding the patient's health and treatment status;
  * enable the collection of data relating to episodes of fever and/or acute pain (Fever Diary, Pain Diary, and Other Events/Symptoms Diary);
  * manage the Fever Diary and Pain Diary, therapy planning, and therapeutic reconnaissance (for appropriateness purposes).

SUMMARY:
FEVER is a single-center, prospective, open-label, pre-market, pivotal, single-arm study aimed at demonstrating how the use of an algorithm integrated with a Class I Medical Device (Puntofarma®), which is made available through a downloadable mobile phone app, can, given specific input, improve the appropriateness and adherence to therapy for the management of fever and pain in children between 3 months and 1 day and 5 years of age.

100 patients are expected to be enrolled, equally distributed between febrile patients (50%) and patients with acute pain (50%). Patients admitted to the Regional Pediatric Emergency Department of the Meyer IRCCS Hospital in the presence of a feverish episode and/or acute pain will be enrolled upon discharge.

The study will last a total of 8 months (Jan - Aug 2026), with enrollment expected by Jan 2026. Each patient will be involved in the study for a maximum of 7 days from enrollment, during which they will use the mobile app. Participation in the study will conclude by the seventh day of use of the app, with the completion of a satisfaction questionnaire.

DETAILED DESCRIPTION:
FEVER is a single-center, prospective, open-label, pre-market, pivotal, single-arm study aimed at demonstrating how the use of an algorithm integrated with a medical device (Puntofarma®), given specific input, can improve the appropriateness and adherence to pharmacological therapy with paracetamol for the management of fever and acute pain in patients between 3 months and 1 day and 5 years of age. The algorithm for digital pharmacological support was developed based on therapeutic guidelines.

The study lasts seven days from the date of enrollment of the individual patient.

Upon admission to the emergency room for an episode of fever and/or acute pain, provided that all eligibility criteria are met, and following receipt of signed informed consent, the investigator will propose the study to the patient's family members or caregivers. The patient will be managed according to clinical standards regarding the presenting condition. Participation in the study, or refusal, will not result in any changes to the flow or management of the patient as required by the current clinical condition or current standards.The study will begin immediately upon the patient's discharge from the emergency room.

After signing the informed consent form, the patient and caregiver will be enrolled in the study and registered in the Puntofarma® system, resulting in the issuance of a unique code.

No personal data of the patient and/or caregiver will be recorded on the device. At the same time, each enrolled patient will be issued a PIN code through which the caregiver will be able to register in the digital application and begin using the algorithm from their mobile/digital device. Caregivers will be asked to enter the information in the application necessary for the algorithm to calculate the recommended dose of paracetamol. The application, which can be downloaded to a mobile phone, is used to verify adherence to the antipyretic therapy suggested by the algorithm, which is based on the guidelines for the management of fever and acute pain in children.

No follow-up visits, tests, or additional services are scheduled during the seven-day investigation. Seven days after patient enrollment, at the conclusion of the study, the parent/caregiver will be given a questionnaire (also via the app) to assess the usability and caregiver satisfaction with the use of the app.

The app includes an optional diary, relating to fever, pain, or other symptoms/events, in which it is also possible to record additional information and to report adverse events or device defects.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, male or female, between 3 months and 1 day and 5 years of age, who have a fever and are prescribed paracetamol, or who have already received a prescription for an antipyretic from an outside physician before accessing the emergency room.
* Pediatric patients, male or female, between 3 months and 1 day and 5 years of age, who have acute pain and are prescribed paracetamol, or who have already received a prescription for an analgesic from an outside physician before accessing the emergency room.
* Pediatric patients whose caregivers have knowledge of the Italian language.
* Pediatric patients whose caregivers have access to the internet and have a smartphone that is either the latest generation or no older than five years.

Exclusion Criteria:

* Pediatric patients, male or female, aged less than 3 months and over 5 years.
* Pediatric patients who have experienced adverse reactions or contraindications to paracetamol administration.
* Pediatric patients whose caregivers have little or no knowledge of the Italian language.
* Pediatric patients whose caregivers do not have internet access or do not have a latest-generation smartphone or, in any case, one no older than five years.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of adherence to the prescribed dosage of paracetamol during the treatment cycle. | 8 days of treatment
  Measurement of adherence to the prescribed dosage of paracetamol during the treatment cycle.

SECONDARY OUTCOMES:
Evaluation of the consistency of the timing of paracetamol administration during the treatment period | 8 days of intervention
  Evaluation of the consistency of the timing of paracetamol administration during the treatment period
Digital app usage rate: Percentage of parents/caregivers using the digital app | 8 days of intervention
  Digital app usage rate:
  Percentage of parents/caregivers using the digital app
Number (%) of patients taking ibuprofen | 8 days of intervention
  Number (%) of patients taking ibuprofen
Caregiver satisfaction | 8 days of intervention
  Satisfaction level using a rating scale. Caregiver satisfaction:
  Measured using a structured questionnaire/Likert scale to evaluate the user experience and perceived usefulness of the application

CONTACTS AND LOCATIONS:
Overall Officials: Niccolò Parri, MD, Pediatric Emergency, Principal Investigator — Meyer University Children's Hospital Florence, Department of Emergency Medicine and Trauma Center, ITALY
Locations (1):
- Meyer University Children's Hospital Florence, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Under review by the Sponsor